CLINICAL TRIAL: NCT01259401
Title: Treating Sleep Problems in VA Adult Day Health Care
Acronym: HERO-ADHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E7037-R
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Insomnia; Sleep Disorders
Keywords: Sleep; Rehabilitation; Behavior therapy; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIP group (Experimental): The Sleep Intervention Program group received a sleep education program based on behavioral principles, delivered in 4 individual sessions carried out within the Adult Day Health Care program.
  Interventions: Behavioral: Sleep Intervention Program
- Control group (Active Comparator): The Control group received basic sleep education, delivered in 4 individual sessions carried out within the Adult Day Health Care
  Interventions: Behavioral: Sleep Education control

INTERVENTIONS:
Behavioral: Sleep Intervention Program — Sessions focused on: 1) sleep consolidation and sleep schedule optimization, 2) sleep hygiene education, 3) cognitive therapy, and 4) maintenance of sleep improvements and coping with future bouts of insomnia.
  Arms: SIP group
Behavioral: Sleep Education control — During sessions, participants reviewed two educational brochures that focused on changes in sleep with age and sleep hygiene education.
  Arms: Control group

SUMMARY:
The Veterans Millennium Health Care and Benefits Act (Millennium Act) of 1999 mandated the Department of Veterans Affairs (VA) to provide non-institutional long-term care to veterans. Adult Day Health Care (ADHC) is a key component of that spectrum of long-term care services. Veterans in ADHC commonly suffer from limited poor functioning, depression, cognitive problems and low quality of life. These factors can lead to continued deterioration in functioning, loss of independence, hospitalizations, nursing home placement and death. Sleep disruption is associated with depression, low quality of life, functional decline, nursing home placement, and death among older people. Sleep disturbance is common among ADHC patients, it is not addressed within routine clinical care, and treatment may be limited to medications. Studies show that untreated insomnia and medications for insomnia can increase risk of falls and other health events among older persons. On the other hand, non-medication treatments for sleep do not show these problems. These treatments have been shown to be effective in other studies. The goal of this study is to test non-medication treatments to improve sleep among older Veterans with insomnia in a VA ADHC program. The study design will facilitate translation into routine care and application in other similar VA programs.

DETAILED DESCRIPTION:
The Veterans Millennium Health Care and Benefits Act (Millennium Act) of 1999 mandated the Department of Veterans Affairs (VA) to provide non-institutional long-term care to veterans. Adult Day Health Care (ADHC) is a key component of that spectrum of long-term care services. ADHC provides health maintenance, rehabilitation services and socialization in a group setting during daytime hours. Veterans in ADHC commonly suffer from limited physical functioning, depression, cognitive difficulties and low quality of life. These factors increase the likelihood of continued deterioration in functioning, loss of independence, hospitalizations, nursing home placement and death. Previous studies, including our own work, have demonstrated that sleep disruption is associated with depression, low quality of life, functional decline, nursing home placement, and death among older people. The investigators have found that sleep disturbance is common among ADHC patients, it is not addressed within routine clinical care, and treatment is commonly limited to medications (e.g., hypnotics, sedating antidepressants). Numerous studies show that both untreated insomnia and pharmacological treatment of insomnia can be associated with increased risk of falls and other adverse health events among older persons. On the other hand, nonpharmacological interventions on sleep do not show these adverse effects, have been shown to be effective and are associated with improvements in mood, quality of life and health.

The goal of the study was to test the effectiveness of a cognitive-behavioral intervention to improve self-reported and objectively-measured sleep quality among older veterans with insomnia in a VA ADHC program. The intervention program involved a 4-session manualized treatment. This Sleep Intervention Program (SIP) was compared to an active Sleep Education control that also included 4 individual sessions using a randomized trial with 72 veterans. To our knowledge, this study is the first to address the unmet need for non-pharmacological treatment of sleep problems among ADHC patients. The intervention design (e.g., use of a manualized treatment that can be provided by non-psychologists) will facilitate translation into routine care and application in other similar VA programs.

ELIGIBILITY:
Inclusion Criteria:

All of the following:

* ADHC program participant
* Age >= 60 years
* Ability to communicate verbally

Exclusion Criteria:

One or more of the following:

* Significant cognitive impairment (Mini Mental State Examination score<20)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Martin, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

REFERENCES:
- [Result] Song Y, Dzierzewski JM, Fung CH, Rodriguez JC, Jouldjian S, Mitchell MN, Josephson KR, Alessi CA, Martin JL. Association Between Sleep and Physical Function in Older Veterans in an Adult Day Healthcare Program. J Am Geriatr Soc. 2015 Aug;63(8):1622-7. doi: 10.1111/jgs.13527. Epub 2015 Jul 22. PMID 26200520
- [Derived] Martin JL, Song Y, Hughes J, Jouldjian S, Dzierzewski JM, Fung CH, Rodriguez Tapia JC, Mitchell MN, Alessi CA. A Four-Session Sleep Intervention Program Improves Sleep for Older Adult Day Health Care Participants: Results of a Randomized Controlled Trial. Sleep. 2017 Aug 1;40(8):zsx079. doi: 10.1093/sleep/zsx079. PMID 28482053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans enrolled in the ADHC program for at least one month were screened for study eligibility criteria (i.e., the ability to understand screening items and to communicate during the screening process. If the individual was interested, written informed consent was obtained.
Pre-assignment Details: A total of 72 participants were enrolled into the study. After baseline assessment, 30 participants were not eligible for randomization: too cognitive impaired to participate (13); medical or behavioral issue (n=6); no longer met criteria for insomnia (n=3); discharged from ADHC (n=4); refused randomization (n=2); withdrew (n=2).
Groups:
- SIP Group: The SIP group received a sleep education program based on behavioral principles, delivered in 4 individual sessions carried out within the Adult Day Health Care program.
  Sleep Intervention Program: Sessions focused on: 1) sleep consolidation and sleep schedule optimization, 2) sleep hygiene education, 3) cognitive therapy, and 4) maintenance of sleep improvements and coping with future bouts of insomnia.
- Control Group: The control group received basic sleep education, delivered in 4 individual sessions carried out within the Adult Day Health Care
  Sleep Education control: During sessions, participants reviewd two educational brochures that focused on changes in sleep with age and sleep hygiene education.
Period: End of 4-week Intervention
Arm/Group | SIP Group | Control Group
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: 4-month Follow-up
Arm/Group | SIP Group | Control Group
Started | 21 | 21
Completed | 21 | 19
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIP Group | Control Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (10.2) | 76.4 (9.9) | 77.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 18 | 21 | 39
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 17 | 30
  Non-white | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Percentage of time asleep while in bed estimated by actigraphy
Time Frame: End of 4-week intervention
Population: Two SIP subjects had missing data for this variable.
Measure: Mean (95% Confidence Interval); unit: percentage of time in bed spent asleep
Arm/Group | SIP Group | Control Group
Number analyzed (Participants) | 19 | 21
percentage of time in bed spent asleep | 86.6 [84.3 to 88.8] | 83.3 [81.2 to 85.4]
Statistical Analysis 1: Comparison: SIP Group vs Control Group; Test type: Superiority or Other; p = .04, ANCOVA

2. Primary Outcome: Sleep Efficiency
Description: Percentage of time asleep while in bed estimated by actigraphy.
Time Frame: 4-month follow-up
Population: Two SIP subjects had missing data for this variable.
Measure: Mean (95% Confidence Interval); unit: percentage of time in bed asleep
Arm/Group | SIP Group | Control Group
Number analyzed (Participants) | 19 | 19
percentage of time in bed asleep | 85.3 [82.5 to 88.1] | 81.5 [78.7 to 84.3]
Statistical Analysis 1: Comparison: SIP Group vs Control Group; Test type: Superiority or Other; p = .061, ANCOVA

ADVERSE EVENTS:
Time Frame: Four months
Arm/Group | SIP Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SIP Group (N=21) | Control Group (N=21)
Wrist abrasion from actigraph (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Small sample size; predominantly male study sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes